CLINICAL TRIAL: NCT02243631
Title: ANK-dependent ATP Efflux Causes Calcium Pyrophosphate Deposition in Cartilage
Brief Title: Effect of Probenecid on Synovial Fluid ATP Levels in CPPD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMMA-022-13F
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Results first posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Calcium Pyrophosphate Deposition Disease
Keywords: ATP; Probenecid; Chondrocalcinosis
MeSH Terms: conditions — Chondrocalcinosis | interventions — Probenecid; Uricosuric Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probenecid (Experimental): These patients will receive 5 days of probenecid.
  Interventions: Drug: Probenecid
- No intervention (No Intervention): These patients will receive no intervention.

INTERVENTIONS:
Drug: Probenecid — Treatment
  Other Names: uricosuric
  Arms: Probenecid

SUMMARY:
This study will investigate the hypothesis that probenecid, a medication currently used for gout, reduces levels of ATP in the joint fluid of patients with calcium pyrophosphate deposition disease (CPPD), another common type of crystal-related arthritis. There is good evidence that CPPD results from an excess of ATP in joints. The investigators will measure levels of ATP in joint fluid before and after 5 days of treatment with probenecid. This study will serve to rationalize larger studies of probenecid in CPPD.

DETAILED DESCRIPTION:
Objective: The objective of this study is to determine whether pharmacologic doses of the drug probenecid significantly decrease ATP and inorganic pyrophosphate (PPi) levels in the synovial fluid of patients with calcium pyrophosphate deposition disease (CPPD). The investigators have considerable evidence that synovial fluid ATP levels are high in patients with this disease and these high levels lead to calcium pyrophosphate (CPP) crystal formation which then produces acute and chronic arthritis. The investigators have identified the transmembrane protein known as ANK as the chief regulator of ATP levels in and around cartilage. Probenecid blocks function of ANK in vitro. The purpose of this study is to determine if probenecid used at normal doses are sufficient to block ANK function in vivo and whether this results in reduced ATP and PPi levels in synovial fluid.

Research design: This is a randomized un-controlled trial of probenecid vs. no drug in patients with a joint effusion and known CPPD.

Methodology: Power analysis based on an 80% chance to show a 20% difference in ATP levels in the treatment group resulted in a sample size of 20 patients in each group. Patients with known CPPD and a joint effusion will have an arthrocentesis to remove 2 ml of synovial fluid from their joint. Fluid will be sent to the investigators' research laboratory and ATP and PPi levels will be measured. Patients will be randomized to treatment with 2 grams/day of probenecid or no therapy. After 5 days, the remainder of the joint fluid will be removed and tested for ATP and PPi levels. The investigators will compare differences in ATP and PPi levels in the probenecid treated and the untreated group.

ELIGIBILITY:
Inclusion Criteria:

* Age >21 years,
* CPPD diagnosed by Ryan /McCarty criteria
* Joint effusion in a shoulder or knee

Exclusion Criteria:

* Inability to sign informed consent
* Age <21 years
* History of renal stones
* Significant renal dysfunction (CKD >stage 2)
* Blood dyscrasias
* Current use of drugs which interact with probenecid
* Concurrent gout
* Active infection, including bacteremia and overlying cellulitis
* Recent joint trauma
* Intra-articular corticosteroids in the affected joint within three months

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann K Rosenthal, MD, Principal Investigator — Clement J. Zablocki VA Medical Center, Milwaukee, WI
Locations (1):
- Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Probenecid | No Intervention
Started | 3 | 5
Completed | 3 | 4
Not Completed | 0 | 1
Not completed — no synovial fluid on second aspirate | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probenecid | No Intervention | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.6 (12.3) | 68.4 (10.4) | 71.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 5 | 8
ATP levels in synovial fluid at day 0 [Mean (Standard Deviation); unit: nanomoles/ml] | 1.2 (0.9) | 4.5 (6.7) | 2.85 (2.33)

OUTCOME MEASURES:

1. Primary Outcome: ATP Levels in Synovial Fluid
Description: The investigators will measure levels of ATP in synovial fluid from patients with CPPD before and after treatment with probenecid compared to patients receiving no therapy. ATP levels are measured with a standard bioluminescent assay.
Time Frame: 5 days
Population: Two subjects ( one in probenecid and one in no intervention group) had no measurable ATP on the second aspirate, and one subject in the no intervention group did not have any synovial fluid on the second visit.
Measure: Mean (Standard Deviation); unit: nanomoles/ml
Groups:
- Probenecid: probenecid group after 5 days of drug
- no Intervention: no intervention after 5 days
Arm/Group | Probenecid | no Intervention
Number analyzed (Participants) | 2 | 3
nanomoles/ml | 4.4 (2.5) | 31.4 (56.6)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Probenecid | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT02243631/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT02243631/ICF_001.pdf